CLINICAL TRIAL: NCT04561726
Title: The Effects of Connective Tissue Manipulation on Balance and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bahçeşehir University (Other); Yeditepe University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 37068608-6100-15-1477
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Connective tissue massage; Connective Tissue Manipulation; Proprioception; Postural Balance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The sample size was calculated before starting to study by the G*Power 3.1.9.2. In order to find a meaningful difference between the pre-treatment and post-treatment Biodex Balance System (BBS) measurements, study group should include at least 18 individuals when the type I error was 0.5 and 95% power value (1-β = 0.95). Considering the data loss that may occur during the study period, 20 volunteers were planned for each group (40 voluntary university students in total).
Who Masked: Participant
Masking Description: The volunteers were numbered according to the order of their application. At the end of the applications, small papers were numbered from 1 to 40, and among these papers, the first 20 people selected by the lottery method were included in the study group, and the rest were included in the exercise group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): All of the 20 participants in the study group were asked to do the given 11 home exercises (balance, stretching and strengthening exercises) twice a week for 6 weeks. The exercises were progressed day by day. All of the exercises were taught in the first assessment day, after the all measurements collected. All participants were controlled every week by social media and face-to-face conversations.
  Additionally, CTM was applied to the volunteers in study group for 6 weeks, 2 sessions in a week.CTM applied to lumbosacral area (basic region), lower toracal, scapular, interscapular and cervical regions, respectively.
  Interventions: Other: Connective Tissue Manipulation; Other: Exercise
- Exercise Group (Active Comparator): All of the 20 participants in the exercise group were asked to do the given 11 home exercises (balance, stretching and strengthening exercises) twice a week for 6 weeks. The exercises were progressed day by day. All of the exercises were taught in the first assessment day, after the all measurements collected. All participants were controlled every week by social media and face-to-face conversations.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Connective Tissue Manipulation — Connective tissue manipulation is a soft tissue manipulative technique and also a reflex therapy which is characterized by localised and specific strokes performed in where the fascia is superficial or palpable. A shear force is created between the skin-underlying fascia or dermis-hypodermis and angulatory force is applied to the collagen fibers to produce reflex and mechanical effects.
  Other Names: Connective Tissue Massage
  Arms: Study Group
Other: Exercise — The purpose of the given home exercises is to increase motor ability in activities such as standing, walking and posture, to increase muscle strength and also to elongate muscles. Exercises progressed day by day according to the adaptation of the motor system and muscle strength to the exercises.

SUMMARY:
There are various exercises and manual techniques to improve balance and proprioception. Most of these manual therapy techniques are mobilization, manipulation, post-isometric relaxation, myofascial relaxation and traction massage. At the same time, it has been observed that many parameters such as range of motion, tissue tension, wound healing process and pain perception were examined in the studies in the literature, but the effects of CTM on balance and proprioception have not been investigated.

The aim of the study was to investigate the effects of CTM on balance and proprioception among healthy individuals. 40 volunteers studying in Bahcesehir University were divided into 1) exercise and 2) study (CTM with exercise) groups equally. Both exercise and study groups were instructed to perform home exercises for 2 sessions in a week for 6 weeks (12 sessions in total). Additionally, CTM was applied to the volunteers in study group for 6 weeks, 2 sessions in a week. CTM applied to the lower and the upper back, and also neck.

Balance, cervical and lumbar proprioception was measured to understand the effectiveness of the CTM. Biodex Balance System was used for evaluation of static and dynamic balance. The cervical proprioception was measured by using a cervical range of motion (CROM) device while lumbar proprioception was measured by StabilizerTM Pressure Biofeedback Unit. Additionally, heart rate and blood pressure were measured by M3 Comfort Digital blood Pressure Monitor. All measurements applied at the beginnig and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being voluntary
* Being healthy enough not to be constantly under the control of a health institution
* Being over 18 years old

Exclusion Criteria:

* Having neurological or orthopedic problems that can influence lower extremity functions and balance,
* Having any kind of vestibular system problems (Vertigo, Meniere etc.)
* Having a surgery from lumbar, thoracic or/and cervical regions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System (BBS) | 10 minutes
  The BBS, which consists of a monitor connected multi-axis platform, objectively measures static and dynamic balance and records measurement results as degrees for three directions: medial lateral stability index, anterior-posterior stability index, and overall stability index. These indices show the fluctuations around the zero point. The mobility of the platform can be adjusted allowing the static and dynamic balance to be measured.
  Postural Stability Protocol has been selected from 5 test protocols of BBS. In this protocol, the aim is to try to match the ball seen on the screen to the midpoint of the ring shaped screen by transferring the weight on the platform. Firstly, static platform were used and volunteers stand on both foot, then on right and left foot. Then, the same measurements were repeated on dynamic platform which is level 4 out of 8. Each measurement was tested in 3 repetitions. Mean of these repetitions were noted as the score of that measurement.

SECONDARY OUTCOMES:
Cervical Range of Motion Tester (C-ROM) | 10 minutes
  It is glasses-shaped measurement device which indicate the position of the head and consist of two inclinometers which are in sagittal and frontal planes.
  To assess cervical proprioception, flexion and right and left lateral flexion were chosen. When they put on the CROM, we asked them to bend the head forward and we stopped them when they reached 30 degrees and asked them to feel the amount of movement and muscle tension. We repeated the procedure 3 times with eyes open and 3 times with eyes closed. Then we asked the volunteers to flex their heads three times and stop when they thought they reached 30 degrees. Average of each flexion degrees that they stopped was noted and the deviation from the target angle was calculated as score.
  Then the same procedure was repeated for right and left lateral flexion.
Stabilizer Pressure Biofeedback Unit (SPBU) | 5 minutes
  SPBU consists of three-chamber pressure cell connected to gauge and inflation bulb. It is used for the strengthening of the abdominal and erector muscles or teaching the stabilization exercises. In our study, it was used for to measure the ability of the person to return to the pressure level which is taught before. Volunteers were in hook-lying position. They were asked to perform posterior pelvic tilt and the pressure cell was inflated to 40 mmHg. Then, they were asked to relax. Later, the posterior pelvic tilt was performed 3 times with the eyes open and 3 times with the eyes closed so that the volunteers could feel the amount of contraction in the muscles at 40mmHg. Then the test began. As in the trials, the volunteers perform posterior pelvic tilt with eyes open and eyes closed (3 times each) and said "I feel this is 40mmHg" when they thought they reached 40mmHg. The deviation from the target pressure was calculated and averages of 3 measurements were recorded as score.
M3 Comfort Digital Blood Pressure Monitor | 2 minutes
  It is used to measure heart rate and blood pressure. The cuff was placed on the arm in relation to brachial artery. Volunteers were informed about avoiding exercise and not eating or drinking half an hour before blood pressure measurement. It was noted that the clothing was not squeezing the arm. The volunteers were positioned on a chair with back support, both feet on the floor and the upper arm supported at the level of the heart and were asked not to contract any muscle of upper arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No